CLINICAL TRIAL: NCT07096128
Title: A Phase I Study to Assess the Safety, Tolerability, Radiation Dosimetry and Efficacy of [177Lu] Lu-PSMA-XT in Patients With Metastatic Prostate Cancer
Brief Title: A Study of [177Lu] Lu-PSMA-XT Injection in Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jinming Zhang (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor-Investigator, Jinming Zhang, PI, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-XTR021-1-03
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: mCRPC
Keywords: mCRPC; 177Lu; PSMA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu-PSMA-XT (Experimental): [177Lu]Lu-PSMA-XT is a radioligand therapy that delivers beta-particle radiation to PSMA-expressing cells
  Interventions: Drug: [177Lu]Lu-PSMA-XT

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA-XT — [177Lu]Lu-PSMA-XT is a radioligand therapy that delivers beta-particle radiation to PSMA-expressing cells.

SUMMARY:
This was a multicenter, open-label, phase I study to evaluate the safety, tolerability, radiation dosimetry and efficacy of [177Lu] Lu-PSMA-XT injection in patients with metastatic prostate cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and sign an approved informed consent form (ICF).
2. Patients must be >= 18 and <＝80 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Patients must have a life expectancy >6 months.
5. Patients must have histological, pathological, and/or cytological confirmation of prostate cancer.
6. Patients must be PSMA Positron Emission Tomography (PET)/Computed Tomography (CT) scan positive。
7. Patients must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
8. Patients must have received at least one NAAD (such as enzalutamide and/or abiraterone)； patients must have been previously treated undergone at least 1-2 prior taxane-based chemotherapy regimens or be unsuitable for taxane therapy (unsuitability includes contraindications, investigator-determined ineligibility, or patient refusal) in mCRPC stage.
9. Patients must have progressive mCRPC.
10. Patients must have adequate organ function。
11. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, Intra-uterine device（IUD）,etc., during treatment and within 6 months of the last use of the trial drug.

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months of enrollment: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed.
2. Known other malignancies.
3. Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy within 28 days prior to day of enrollment.
4. Known hypersensitivity to the components of the study therapy or its analogs.
5. A superscan as seen in the baseline bone scan.
6. Patients with a history of Central Nervous System (CNS) metastases.
7. Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, or other severe complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
1.Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, assessed up to 2 years
  To evaluate the safety and tolerability of [177Lu]Lu-PSMA-XT Injection assessed from the number and incidence of patients with adverse events using CTCAE v5.0 and physical examination, electrocardiogram and laboratory abnormality, etc.
Dose-limiting toxicity（DLT） | Through study completion, assessed up to 2 years
  Incidence and severity of dose-limiting toxicities.
Whole body and organ uptake of [177Lu]Lu-PSMA-XT Injection | From the first subject enrolled to one week after the last subject completed the first dosing,assessed up to approximately 12 months
  Quantitate the absorbed radiation doses (expressed as Gy/MBq) of administered [177Lu]Lu-PSMA-XT to kidneys, liver, lungs, spleen, bone/red marrow and salivary glands.

SECONDARY OUTCOMES:
Best Percentage Change From Baseline in Prostate-specific Antigen (PSA) Level(PCWG3) | Through study completion, assessed up to 2 years.
  Best percentage change from baseline in PSA level was defined as the maximum percent decrease at any time post-baseline.
Prostate-specific Antigen 50 (PSA50) Response | Through study completion, assessed up to 2 years.
  PSA50 response was defined as the proportion of participants who had a >= 50% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.
Time to PSA progression | Through study completion, assessed up to 2 years.
  PSA progression was defined as: 1) Where a decline from baseline was documented, date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained at least 3 weeks later. Rises in PSA within the first 12 weeks of the date of first dose were ignored; 2) Where no decline from baseline was documented, PSA progression was defined as a >= 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 weeks from the date of first dose (without confirmation) as specified in the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines.
Radiographic Progression-free Survival (rPFS) | Through study completion, assessed up to 2 years.
  Radiographic progression-free survival (rPFS) was defined as the time (in months) from the date of enrollment to the date of radiographic disease progression per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria or death due to any cause.
Overall Response Rate (ORR) | Through study completion, assessed up to 2 years.
  Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline.
Duration of Response (DOR) | Through study completion, assessed up to 2 years.
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause .
Disease Control Rate (DCR) | Through study completion, assessed up to 2 years.
  Disease control rate (DCR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1.
Time to First Symptomatic Skeletal Event (SSE) | Through study completion, assessed up to 2 years.
  Time to first Symptomatic Skeletal Event (SSE) was defined as the time (in months) from the date of enrollment to the date of the SSE or death from any cause. The SSE date was the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Zhang, Principal Investigator — The First Medical Center, Chinese PLA General Hospital
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Mianyang Central Hospital, Beijing, Beijing Municipality
  - The First Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No